CLINICAL TRIAL: NCT01239524
Title: The Significance of Latissimus Dorsi Flap Innervation in Delayed Breast Reconstruction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Responsible Party: Minna Kaariainen/ MD, PhD, Tampere University Hospital, Plastic and Reconstructive surgery department
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R06075
Record Dates: First submitted 2010-11-10; First posted 2010-11-11 (Estimated); Last update posted 2010-11-11 (Estimated); Status verified 2010-11

CONDITIONS: Significance of Latissimus Dorsi Flap Innervation in Delayed Breast Reconstruction
Keywords: breast reconstruction, latissimus dorsi flap, thoracodorsal nerve, skeletal muscle disuse, breast MRI

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DE-group (Other): surgical denervation by excising 1 cm of proximal thoracodorsal nerve
  Interventions: Procedure: denervation of thoracodorsal nerve or saving the nerve
- IN group (Other): thoracodorsal nerve is saved intact
  Interventions: Procedure: denervation of thoracodorsal nerve or saving the nerve

INTERVENTIONS:
Procedure: denervation of thoracodorsal nerve or saving the nerve

SUMMARY:
Breast reconstruction with a pedicled myocutaneous latissimus dorsi (LD) flap is a widely used reconstruction method. It is controversial if surgical denervation by transecting the thoracodorsal nerve should be performed or not. It is assumed that after denervation the latissimus dorsi muscle will significantly atrophy and lose volume. On the other hand discomforting signs and symptoms from muscle contraction are believed to be prevented if flap is denervated. The aim of the study was prospectively evaluate the influence of LD-flap innervation on the functional and aesthetic outcome of delayed breast reconstruction, and to compare the change in muscle structure in breast MRI and histopathology.

ELIGIBILITY:
Inclusion Criteria:

* delayed LD-flap breast reconstruction, no recurrent disease observed

Exclusion Criteria:

* recurrent cancer, partial resection of the breast

Ages: 20 Years to 70 Years | Sex: Female
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)

REFERENCES:
- [Derived] Kaariainen M, Giordano S, Kauhanen S, Helminen M, Kuokkanen H. No need to cut the nerve in LD reconstruction to avoid jumping of the breast: a prospective randomized study. J Plast Reconstr Aesthet Surg. 2014 Aug;67(8):1106-10. doi: 10.1016/j.bjps.2014.04.029. Epub 2014 May 13. PMID 24933238
- [Derived] Kaariainen M, Giordano S, Kauhanen S, Laaperi AL, Mattila P, Helminen M, Kalimo H, Kuokkanen H. The significance of latissimus dorsi flap innervation in delayed breast reconstruction: a prospective randomized study-magnetic resonance imaging and histologic findings. Plast Reconstr Surg. 2011 Dec;128(6):637e-645e. doi: 10.1097/PRS.0b013e318230c544. PMID 22094764